CLINICAL TRIAL: NCT00115778
Title: IVIG for Acquired Immunodeficiency in Lung Transplant Patients
Brief Title: Intravenous Immunoglobulin (IVIG) in Lung Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Grifols Therapeutics LLC (Industry)
Responsible Party: Principal Investigator, Selim Arcasoy, Dickinson W. Richards, Jr. Professor of Medicine (in Pediatrics) at the Columbia University Medical Center, Dept of Medicine Pulmonary, Columbia University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AAAB0431
Record Dates: First submitted 2005-06-26; First posted 2005-06-27 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Hypogammaglobulinemia; Lung Transplantation
Keywords: Hypogammaglobulinemia; Lung Transplantation
MeSH Terms: conditions — Agammaglobulinemia | interventions — Immunoglobulins, Intravenous; gamma-Globulins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- First IVIG, then Placebo (Experimental): Study participants will receive three doses of IVIG given four weeks apart over 12 weeks followed by a twelve-week washout and then three doses of placebo over 12 weeks.
  Interventions: Drug: IVIG; Other: Placebo
- First Placebo, then IVIG (Experimental): Study participants will receive three doses of 0.1% albumin solution (placebo) given four weeks apart over 12 weeks followed by a twelve-week washout and then three doses of IVIG over 12 weeks.
  Interventions: Drug: IVIG; Other: Placebo

INTERVENTIONS:
Drug: IVIG — 10% Caprylate/Chromatography Purified Intravenous Immunoglobulin 400 mg/kg IV every 4 weeks
  Other Names: Immune globulin intravenous; Gamunex; Intravenous immunoglobulin
Other: Placebo — 0.1% Albumin in an equal volume to the investigational product

SUMMARY:
The purpose of this study is to determine if intravenous immunoglobulin (IVIG) can prevent bacterial infections in lung transplant patients with low serum levels of immunoglobulin.

DETAILED DESCRIPTION:
An increased risk of infection despite intensive antimicrobial prophylaxis is a well-recognized complication of lung transplantation. Recent evidence suggests that immunosuppressive therapy after solid organ transplantation may lead to humoral immunodeficiency due to hypogammaglobulinemia (HGG). In lung transplant recipients with HGG, IVIG therapy offers the potential to significantly decrease the incidence and severity of infections, thereby reducing morbidity and potentially mortality.

Comparison: The investigators are conducting a randomized clinical trial of IVIG versus placebo for lung transplant patients with severe HGG to see if IVIG decreases the number of bacterial infections in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Lung transplant recipients > 3 months after transplant surgery
* Immunoglobulin G (IgG) < 500 mg/dL
* Stable medical regimen

Exclusion Criteria:

* Acute rejection
* Active infection
* Contraindication to IVIG
* Pregnancy
* Recent thrombotic event

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2005-06; Primary Completion 2009-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Selim M Arcasoy, M.D., Principal Investigator — Columbia University
Locations (1):
- New York Presbyterian Hospital Lung Transplant Program, New York, New York, United States

REFERENCES:
- [Result] Lederer DJ, Philip N, Rybak D, Arcasoy SM, Kawut SM. Intravenous immunoglobulin for hypogammaglobulinemia after lung transplantation: a randomized crossover trial. PLoS One. 2014 Aug 4;9(8):e103908. doi: 10.1371/journal.pone.0103908. eCollection 2014. PMID 25090414

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eleven subjects were eligible and randomized, and 10 completed all study assessments. One subject discontinued the interventions because of inability to comply with the schedule of study visits. 10 subjects are needed to detect a reduction in the mean number of bacterial infections/patient by one standard deviation over three months with 80% power.
Groups:
- Group 1: Placebo Then IVIG: Study participants consented to receive three doses of 0.1% albumin solution (placebo) given four weeks apart over 12 weeks (period 1) followed by a twelve-week washout and then three doses of IVIG over 12 weeks (period 2).
  Period 1 (12 weeks) Washout period (12 weeks) Period 2 (12 weeks)
  Analysis: modified intention-to-treat
- Group: 2 IVIG Then Placebo: Study participants consented to receive three doses of IVIG given four weeks apart over 12 weeks (period 1) followed by a twelve-week washout and then three doses of placebo over 12 weeks (period 2).
  Period 1 (12 weeks) Washout period (12 weeks) Period 2 (12 weeks)
  Analysis: modified intention-to-treat
Period: Overall Study
Arm/Group | Group 1: Placebo Then IVIG | Group: 2 IVIG Then Placebo
Started | 6 | 5
Completed | 6 | 4
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Study participants consented to receive three doses of IVIG (or 0.1% albumin solution (placebo)) given four weeks apart followed by a twelve-week washout and then three doses of placebo (or IVIG).
Arm/Group | All Participants
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 60 [28 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Clinically Diagnosed Bacterial Infections During the Treatment Period
Description: The number of events occurring during the treatment period. The data will be presented by the occurrence during the IVIG vs. the placebo treatment period, regardless of the order that the treatment was received. Only the clinically diagnosed bacterial infections will be counted.
Time Frame: 3 month
Population: The crossover design, in which each subject serves as his or her own control, allows sufficient power for the detection of a clinically significant effect of IVIG with only a small number of patients. A sample size of 10 patients in a crossover trial has more power to detect differences than double the sample size using a parallel design.
Measure: Number; unit: Infections
Groups:
- Participants Receiving IVIG During Period 1 or Period 2: Study participants received three doses of IVIG first (Period 1) or second (Period 2 - after a twelve-week washout).
- Participants Receiving Placebo During Period 1 or Period 2: Study participants received three doses of placebo first (Period 1) or second (Period 2 - after a twelve-week washout).
Arm/Group | Participants Receiving IVIG During Period 1 or Period 2 | Participants Receiving Placebo During Period 1 or Period 2
Number analyzed (Participants) | 10 | 10
Infections | 3 | 1

2. Secondary Outcome: Number of Clinically Diagnosed Viral Infections
Description: This is to measure the effect of IVIG on viral infections.
Time Frame: 3 month
Measure: Number; unit: Number of Infections
Arm/Group | Participants Receiving IVIG During Period 1 or Period 2 | Participants Receiving Placebo During Period 1 or Period 2
Number analyzed (Participants) | 10 | 10
Number of Infections | 2 | 2

3. Secondary Outcome: Number of Hospital Admissions
Description: This is to measure the effect of IVIG on hospitalizations.
Time Frame: 3 month
Measure: Number; unit: Admissions
Arm/Group | Participants Receiving IVIG During Period 1 or Period 2 | Participants Receiving Placebo During Period 1 or Period 2
Number analyzed (Participants) | 10 | 10
Admissions | 3 | 1

4. Secondary Outcome: Number of Antibiotic Initiation
Description: This is to measure the effect of IVIG on the use of antibiotics.
Time Frame: 3 month
Measure: Number; unit: Uses of antibiotics
Arm/Group | Participants Receiving IVIG During Period 1 or Period 2 | Participants Receiving Placebo During Period 1 or Period 2
Number analyzed (Participants) | 10 | 10
Uses of antibiotics | 9 | 8

5. Secondary Outcome: Number of Clinically Diagnosed Fungal Infection
Description: This is to measure the effect of IVIG on fungal infections.
Time Frame: 3 months
Measure: Number; unit: Infections
Arm/Group | Participants Receiving IVIG During Period 1 or Period 2 | Participants Receiving Placebo During Period 1 or Period 2
Number analyzed (Participants) | 10 | 10
Infections | 2 | 0

6. Secondary Outcome: Number of Lymphocytic Bronchiolitis
Description: This is to measure the effect of IVIG on lung function.
Time Frame: 3 months
Measure: Number; unit: Instances of bronchiolitis
Arm/Group | Participants Receiving IVIG During Period 1 or Period 2 | Participants Receiving Placebo During Period 1 or Period 2
Number analyzed (Participants) | 10 | 10
Instances of bronchiolitis | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Participants Receiving IVIG During Period 1 or Period 2 | Participants Receiving Placebo During Period 1 or Period 2
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 3/10 | 1/10
Other Adverse Events (participants affected / at risk) | 7/10 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Receiving IVIG During Period 1 or Period 2 (N=10) | Participants Receiving Placebo During Period 1 or Period 2 (N=10)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vitreous hemorrhage (Eye disorders) | 1 (1) | 0 (0)
E. coli pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hospital admission for thymoglobulin infusion (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Participants Receiving IVIG During Period 1 or Period 2 (N=10) | Participants Receiving Placebo During Period 1 or Period 2 (N=10)
Fever (General disorders) | 2 | 0
Night sweats (General disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pedal edema (Musculoskeletal and connective tissue disorders) | 0 | 3
Headache (General disorders) | 2 | 3
Stiff neck (Musculoskeletal and connective tissue disorders) | 2 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less